CLINICAL TRIAL: NCT03723616
Title: Exploring Reactions to Health Warnings on Waterpipe Tobacco Ads
Brief Title: Reactions to Warnings on Hookah Ads
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Pro00092330
Record Dates: First submitted 2018-10-26; First posted 2018-10-29 (Actual); Results first posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Reactions to Warnings; Hookah Smoking
Keywords: Hookah; Shisha; Tobacco; Narghile
MeSH Terms: conditions — Water Pipe Smoking

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Social Allure Ads (Active Comparator): Described below is Phase 3. Phase 1 and Phase 2 were small pilots used to inform and select study stimuli. Phase 3 was the larger randomized controlled online trial testing effects of warnings on social allure ads..
  Participants were randomized to one of three health warning label (HWL) arms in a 1:2:2 ratio: 1) ads only, 2) ads with text HWLs only, and 3) ads with text + graphic HWLs. Within the latter two groups, participants were then randomized with equal probability to view HWLs in one of four domains: long- and short-term health events, toxicants, and addiction; participants viewed two HWLs within each domain - there were two HWLs per domain. The text or text + graphic HWLs were placed randomly on two social allure ad themes without replacement. Thus, participants viewed two HWLs within the same domain, with each warning being placed on a different social allure ad. Participants in the ads only arm, only viewed two ads without replacement.
  Interventions: Behavioral: Ads Only; Behavioral: Ads with text-only health warning labels (HWLs); Behavioral: Ads with text + graphic health warning labels (HWLs)
- Product Ads (Active Comparator): Described below is Phase 3. Phase 1 and Phase 2 were small pilots used to inform and select study stimuli. Phase 3 was the larger randomized controlled online trial testing effects of warnings of product ads.
  Participants were first randomized to one of three health warning label (HWL) arms in a 1:2:2 ratio: 1) ads only, 2) ads with text HWLs only, and 3) ads with text + graphic HWLs. Within the latter two groups, participants were then randomized with equal probability to view HWLs in one of four domains: long- and short-term health events, toxicants, and addiction; participants viewed two HWLs within each domain - there were two HWLs per domain. The text or text + graphic HWLs were placed randomly on two ads that represented a flavored tobacco product or a waterpipe apparatus. Thus, participants viewed two HWLs within the same domain, with each warning being placed on a product ad Participants in the ads only arm, only viewed two product ads without replacement.
  Interventions: Behavioral: Ads Only; Behavioral: Ads with text-only health warning labels (HWLs); Behavioral: Ads with text + graphic health warning labels (HWLs)

INTERVENTIONS:
Behavioral: Ads Only — Participants will view 2 ads without replacement.
Behavioral: Ads with text-only health warning labels (HWLs) — Participants will view HWLs in one of four domains: long- and short-term health events, toxicants, and addiction; participants viewed two HWLs within each domain - there were two HWLs per domain. The text HWLs were placed randomly on two ads out of the possible four ad themes without replacement. Thus, participants viewed two HWLs within the same domain, with each warning being placed on a different ad.
Behavioral: Ads with text + graphic health warning labels (HWLs) — Participants will view HWLs in one of four domains: long- and short-term health events, toxicants, and addiction; participants viewed two HWLs within each domain - there were two HWLs per domain. The text + graphic HWLs were placed randomly on two ads out of the possible four ad themes without replacement. Thus, participants viewed two HWLs within the same domain, with each warning being placed on a different ad.

SUMMARY:
The purpose of this study is to help us better understand what kinds of waterpipe tobacco advertisements appeal to young adults as well as to help evaluate and create health warnings that can be placed on waterpipe tobacco advertisements to inform young adults of the risks associated with smoking hookah tobacco.

ELIGIBILITY:
Inclusion Criteria:

* Young adults who are susceptible to or who are current tobacco smokers (which is defined as at least once in the past month, and using hookah tobacco on at least a monthly basis).
* Must have Internet access for Phase 1 and Phase 2 and have a Turkprime account.
* English speaker

Exclusion Criteria:

* Anyone who is not susceptible to waterpipe tobacco smoking or is not a current waterpipe tobacco smoker
* Anyone who does not have Internet access or a Turkprime account

Ages: 18 Years to 34 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 2588 (Actual)
Dates: Start 2018-10-05 (Actual); Primary Completion 2021-03-26 (Actual); Study Completion 2021-03-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Isaac Lipkus, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were randomized to one of three health warning label (HWL) arms in a 1:2:2 ratio: 1) ads only, 2) ads with text HWLs only, and 3) ads with text + graphic HWLs within the Social Allure Ads and Product Ads groups.
Groups:
- Social Allure Ads Only: Behavioral: Ads Only Participants will view 2 ads without replacement.
- Social Allure Ads With Text-only Health Warning Labels (HWLs): Behavioral: Ads with text-only health warning labels (HWLs) Participants will view HWLs in one of four domains: long- and short-term health events, toxicants, and addiction; participants viewed two HWLs within each domain - there were two HWLs per domain. The text HWLs were placed randomly on two ads out of the possible four social allure ad themes without replacement. Thus, participants viewed two HWLs within the same domain, with each warning being placed on a different social allure ad.
- Social Allure Ads With Text + Graphic Health Warning Labels (HWLs): Behavioral: Ads with text + graphic health warning labels (HWLs) Participants will view HWLs in one of four domains: long- and short-term health events, toxicants, and addiction; participants viewed two HWLs within each domain - there were two HWLs per domain. The text + graphic HWLs were placed randomly on two ads out of the possible four social allure ad themes without replacement. Thus, participants viewed two HWLs within the same domain, with each warning being placed on a different social allure ad.
- Product Ads Only: Behavioral: Ads Only Participants will view 2 ads without replacement. Behavioral: Ads with text-only health warning labels (HWLs) Participants will view HWLs in one of four domains: long- and short-term health events, toxicants, and addiction; participants viewed two HWLs within each domain - there were two HWLs per domain. The text HWLs were placed randomly on two ads out of the possible four product ad themes without replacement. Thus, participants viewed two HWLs within the same domain, with each warning being placed on a different product ad.
  Behavioral: Ads with text + graphic health warning labels (HWLs) Participants will view HWLs in one of four domains: long- and short-term health events, toxicants, and addiction; participants viewed two HWLs within each domain - there were two HWLs per domain. The text + graphic HWLs were placed randomly on two ads out of the possible four product ad themes without replacement. Thus, participants viewed two HWLs within the same domain, with each warning being placed on a different product ad.
- Product Ads With Text-only Health Warning Labels (HWLs): Behavioral: Ads with text-only health warning labels (HWLs) Participants will view HWLs in one of four domains: long- and short-term health events, toxicants, and addiction; participants viewed two HWLs within each domain - there were two HWLs per domain. The text HWLs were placed randomly on two ads out of the possible four product ad themes without replacement. Thus, participants viewed two HWLs within the same domain, with each warning being placed on a different product ad.
- Product Ads With Text + Graphic Health Warning Labels (HWLs): Behavioral: Ads with text + graphic health warning labels (HWLs) Participants will view HWLs in one of four domains: long- and short-term health events, toxicants, and addiction; participants viewed two HWLs within each domain - there were two HWLs per domain. The text + graphic HWLs were placed randomly on two ads out of the possible four product ad themes without replacement. Thus, participants viewed two HWLs within the same domain, with each warning being placed on a different product ad.
Period: Overall Study
Arm/Group | Social Allure Ads Only | Social Allure Ads With Text-only Health Warning Labels (HWLs) | Social Allure Ads With Text + Graphic Health Warning Labels (HWLs) | Product Ads Only | Product Ads With Text-only Health Warning Labels (HWLs) | Product Ads With Text + Graphic Health Warning Labels (HWLs)
Started | 317 | 618 | 618 | 207 | 415 | 414
Completed | 300 | 602 | 598 | 201 | 402 | 401
Not Completed | 17 | 16 | 20 | 6 | 13 | 13
Not completed — Attempted to take the survey as both a smoker and a susceptible non-smoker. | 17 | 16 | 20 | 6 | 13 | 13

BASELINE CHARACTERISTICS:
Population: Participants who completed the study. Baseline Characteristics information was collected prior to further stratification into one of three health warning label (HWL) arms in a 1:2:2 ratio: 1) ads only, 2) ads with text HWLs only, and 3) ads with text + graphic HWLs.
Groups:
- Social Allure Ads: Participants were randomized to one of three health warning label (HWL) arms in a 1:2:2 ratio: 1) ads only, 2) ads with text HWLs only, and 3) ads with text + graphic HWLs within the Social Allure Ads group.
  Behavioral: Ads Only Participants will view 2 ads without replacement. Behavioral: Ads with text-only health warning labels (HWLs) Participants will view HWLs in one of four domains: long- and short-term health events, toxicants, and addiction; participants viewed two HWLs within each domain - there were two HWLs per domain. The text HWLs were placed randomly on two ads out of the possible four social allure ad themes without replacement. Thus, participants viewed two HWLs within the same domain, with each warning being placed on a different social allure ad.
  Behavioral: Ads with text + graphic health warning labels (HWLs) Participants will view HWLs in one of four domains: long- and short-term health events, toxicants, and addiction; participants viewed two HWLs within each domain - there were two HWLs per domain. The text + graphic HWLs were placed randomly on two ads out of the possible four social allure ad themes without replacement. Thus, participants viewed two HWLs within the same domain, with each warning being placed on a different social allure ad.
- Product Ads: Participants were randomized to one of three health warning label (HWL) arms in a 1:2:2 ratio: 1) ads only, 2) ads with text HWLs only, and 3) ads with text + graphic HWLs within the Product Ads group.
  Behavioral: Ads Only Participants will view 2 ads without replacement. Behavioral: Ads with text-only health warning labels (HWLs) Participants will view HWLs in one of four domains: long- and short-term health events, toxicants, and addiction; participants viewed two HWLs within each domain - there were two HWLs per domain. The text HWLs were placed randomly on two ads out of the possible four product ad themes without replacement. Thus, participants viewed two HWLs within the same domain, with each warning being placed on a different product ad.
  Behavioral: Ads with text + graphic health warning labels (HWLs) Participants will view HWLs in one of four domains: long- and short-term health events, toxicants, and addiction; participants viewed two HWLs within each domain - there were two HWLs per domain. The text + graphic HWLs were placed randomly on two ads out of the possible four product ad themes without replacement. Thus, participants viewed two HWLs within the same domain, with each warning being placed on a different product ad.
- Total: Total of all reporting groups
Arm/Group | Social Allure Ads | Product Ads | Total
Number analyzed (Participants) | 1500 | 1004 | 2504
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.73 (3.49) | 24.67 (3.46) | 24.71 (3.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 711 | 523 | 1234
  Male | 789 | 481 | 1270
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 247 | 167 | 414
  Not Hispanic or Latino | 1232 | 810 | 2042
  Unknown or Not Reported | 21 | 27 | 48
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 24 | 12 | 36
  Asian | 168 | 104 | 272
  Native Hawaiian or Other Pacific Islander | 5 | 1 | 6
  Black or African American | 165 | 110 | 275
  White | 1010 | 683 | 1693
  Middle Eastern | 17 | 12 | 29
  More than one race | 90 | 55 | 145
  Unknown or Not Reported | 21 | 27 | 48
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 1500 | 1004 | 2504

OUTCOME MEASURES:

1. Primary Outcome: Emotional Reactions to Ads
Description: Participants rated on 7-point bipolar scales the extent each ad made them feel not at all anxious/very anxious, not at all worried/very worried, not at all fearful/very fearful and good /bad. Reported as a composite score created by averaging the items. Mean scores range from 1 to 7 where higher mean values represent more negative emotional reactions to viewing the ad.
Time Frame: up to 45 minutes
Population: Participants who completed the study.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Social Allure Ads Only | Social Allure Ads With Text-only Health Warning Labels (HWLs) | Social Allure Ads With Text + Graphic Health Warning Labels (HWLs) | Product Ads Only | Product Ads With Text-only Health Warning Labels (HWLs) | Product Ads With Text + Graphic Health Warning Labels (HWLs)
Number analyzed (Participants) | 300 | 602 | 598 | 201 | 402 | 401
score on a scale | 2.81 (0.08) | 3.46 (0.06) | 3.74 (0.06) | 2.83 (0.10) | 3.60 (0.07) | 4.03 (0.07)

2. Primary Outcome: Attitudes Toward Waterpipe Tobacco Smoking (WTS) as Measured by Questionnaire
Description: Participant rated on 9-point bipolar scale an ad's portrayal of WTS. The five attributes that tapped cognitions were: safe/unsafe, healthy/unhealthy, useful/useless, harmful/beneficial, and wise/foolish. The five attributes that captured affect were: pleasant/unpleasant, nice/nasty, enjoyable/not enjoyable, satisfying/unsatisfying, gratifying/revolting. Reported as a composite score created by averaging the items. The mean scores could range from 1 to 7 where a higher mean score reflects a more negative attitude towards WTS.
Time Frame: up to 45 minutes
Population: Participants who completed the study.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Social Allure Ads Only | Social Allure Ads With Text-only Health Warning Labels (HWLs) | Social Allure Ads With Text + Graphic Health Warning Labels (HWLs) | Product Ads Only | Product Ads With Text-only Health Warning Labels (HWLs) | Product Ads With Text + Graphic Health Warning Labels (HWLs)
Number analyzed (Participants) | 300 | 602 | 598 | 201 | 402 | 401
score on a scale | 3.79 (0.08) | 4.59 (0.06) | 4.84 (0.06) | 3.87 (0.10) | 4.88 (0.07) | 5.31 (0.07)

3. Primary Outcome: Reactance to Ads
Description: Two items from the University of North Carolina (UNC) short reactance scale were asked from 1=strongly disagree to 7=strongly agree: "This ad is trying to manipulate me", and "This ad annoys me." Reported as a composite score created by averaging the items. Mean scores can range from 1 to 7. A higher mean score reflect higher reactance, meaning that participants felt more reactance (e.g., felt their freedoms were being taken away).
Time Frame: up to 45 minutes
Population: Participants who completed the study.
Measure: Mean (Standard Error); unit: score on a scale
Groups:
- Product Ads Only: Behavioral: Ads Only Participants will view 2 ads without replacement.
Arm/Group | Social Allure Ads Only | Social Allure Ads With Text-only Health Warning Labels (HWLs) | Social Allure Ads With Text + Graphic Health Warning Labels (HWLs) | Product Ads Only | Product Ads With Text-only Health Warning Labels (HWLs) | Product Ads With Text + Graphic Health Warning Labels (HWLs)
Number analyzed (Participants) | 300 | 602 | 598 | 201 | 402 | 401
score on a scale | 3.87 (0.08) | 3.99 (0.06) | 3.91 (0.06) | 3.47 (0.10) | 3.79 (0.07) | 3.82 (0.07)

4. Primary Outcome: Perceived Effectiveness of Health Warnings
Description: Participants used a three-item measure as a gestalt assessment of how well an ad dissuaded WTS. The three items, rated from 1=strongly disagree to 7=strongly agree were: "This ad discourages me from wanting to smoke waterpipe tobacco", "This ad makes me concerned about the health effects of smoking waterpipe tobacco", and "This ad makes smoking waterpipe tobacco seem unpleasant to me". Reported as a composite score created by averaging the items. The mean score could ranged from 1 to 7. A higher mean score reflects that the ad was more effective at dissuading WTS.
Time Frame: up to 45 minutes
Population: Participants who completed the study.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Social Allure Ads Only | Social Allure Ads With Text-only Health Warning Labels (HWLs) | Social Allure Ads With Text + Graphic Health Warning Labels (HWLs) | Product Ads Only | Product Ads With Text-only Health Warning Labels (HWLs) | Product Ads With Text + Graphic Health Warning Labels (HWLs)
Number analyzed (Participants) | 300 | 602 | 598 | 201 | 402 | 401
score on a scale | 2.89 (0.09) | 3.88 (0.06) | 4.13 (0.06) | 3.09 (0.11) | 4.15 (0.07) | 4.46 (0.07)

5. Primary Outcome: Ad Effect on Desire to Smoke
Description: Participants were asked, "To what extent did this ad affect your desire to smoke waterpipe tobacco?" from 1=Reduced my desire a lot to 7=Increased my desire a lot. Mean scores could range from 1 to 7. A higher mean score reflects that the ad increased a participant's desire to smoke waterpipe tobacco.
Time Frame: up to 45 minutes
Population: Participants who completed the study.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Social Allure Ads Only | Social Allure Ads With Text-only Health Warning Labels (HWLs) | Social Allure Ads With Text + Graphic Health Warning Labels (HWLs) | Product Ads Only | Product Ads With Text-only Health Warning Labels (HWLs) | Product Ads With Text + Graphic Health Warning Labels (HWLs)
Number analyzed (Participants) | 300 | 602 | 598 | 201 | 402 | 401
score on a scale | 4.37 (0.08) | 4.07 (0.06) | 3.89 (0.06) | 4.70 (0.10) | 4.03 (0.07) | 3.79 (0.07)

6. Primary Outcome: Ad Effect on Event Participation
Description: Participants who completed the social allure study were asked, "If the activities in the ad were to take place in a location near you, how likely are you to participate in those activities?". Response options were: 1=No chance, 2=Very unlikely, 3=Unlikely, 4=Moderately likely, 5=Likely, 6=Very Likely, and 7=Certain to happen. Mean scores could range from 1 to 7. A higher mean score reflects a higher probability that the participant would participate in the event depicted in the ad.
Time Frame: up to 45 minutes
Population: Only applicable to social allure ad participants who completed the study.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Social Allure Ads Only | Social Allure Ads With Text-only Health Warning Labels (HWLs) | Social Allure Ads With Text + Graphic Health Warning Labels (HWLs) | Product Ads Only | Product Ads With Text-only Health Warning Labels (HWLs) | Product Ads With Text + Graphic Health Warning Labels (HWLs)
Number analyzed (Participants) | 300 | 602 | 598 | 0 | 0 | 0
score on a scale | 3.58 (0.09) | 3.52 (0.06) | 3.43 (0.06) |  |  |

7. Primary Outcome: Ad Effect on Product Purchase
Description: Participants who completed the social allure study were asked, "How likely are you to buy the product in the ad?". Response options were: 1=No chance, 2=Very unlikely, 3=Unlikely, 4=Moderately likely, 5=Likely, 6=Very Likely, and 7=Certain to happen. Means scores could range from 1 to 7. A higher mean score reflects that the study participant would have a higher probability of purchasing the product depicted in the ad.
Time Frame: up to 45 minutes
Population: Only applicable to product ad participants who completed the study.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Social Allure Ads Only | Social Allure Ads With Text-only Health Warning Labels (HWLs) | Social Allure Ads With Text + Graphic Health Warning Labels (HWLs) | Product Ads Only | Product Ads With Text-only Health Warning Labels (HWLs) | Product Ads With Text + Graphic Health Warning Labels (HWLs)
Number analyzed (Participants) | 0 | 0 | 0 | 201 | 402 | 401
score on a scale |  |  |  | 4.04 (0.13) | 3.51 (0.09) | 3.38 (0.09)

8. Secondary Outcome: Perceived Risk as Measured by Questionnaire
Description: Participants responded to three questions tapping perceived personal risk, "What do you think is your chance of getting a serious smoking-related disease in your lifetime, such as cancer, lung disease or heart disease, if you do not quit waterpipe tobacco smoking?" (1=No chance to 7=Certain to happen), "How worried are you about getting a serious smoking-related disease in your lifetime, such as cancer, lung disease, or heart disease, if you do not quit waterpipe tobacco smoking?" (1=Not at all worried to 7=Extremely worried, and "Your 'gut feeling' tells you that you are hurting your health when you smoke waterpipe tobacco?" (1=Strongly disagree to 7=Strongly agree). Reported as a composite score created by averaging the items. Mean scores could range from 1 to 7. A higher mean score reflects a higher overall belief that one is at higher risk for the negative health effects of smoking waterpipe tobacco.
Time Frame: up to 45 minutes
Population: Participants who completed the study.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Social Allure Ads Only | Social Allure Ads With Text-only Health Warning Labels (HWLs) | Social Allure Ads With Text + Graphic Health Warning Labels (HWLs) | Product Ads Only | Product Ads With Text-only Health Warning Labels (HWLs) | Product Ads With Text + Graphic Health Warning Labels (HWLs)
Number analyzed (Participants) | 300 | 602 | 598 | 201 | 402 | 401
score on a scale | 4.71 (0.07) | 4.93 (0.05) | 5.03 (0.05) | 4.73 (0.10) | 4.98 (0.07) | 4.90 (0.07)

9. Secondary Outcome: Global Attitude on Waterpipe Tobacco Smoking (WTS)
Description: Four 7-point bipolar scales tapped views on WTS: negative/positive, dislike/like, bad/good, undesirable/desirable. Reported as a composite score created by averaging the items. The mean scores range from 1 to 7. A higher mean score reflect a more positive overall attitudes towards smoking waterpipe tobacco.
Time Frame: up to 45 minutes
Population: Participants who completed the study.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Social Allure Ads Only | Social Allure Ads With Text-only Health Warning Labels (HWLs) | Social Allure Ads With Text + Graphic Health Warning Labels (HWLs) | Product Ads Only | Product Ads With Text-only Health Warning Labels (HWLs) | Product Ads With Text + Graphic Health Warning Labels (HWLs)
Number analyzed (Participants) | 300 | 602 | 598 | 201 | 402 | 401
score on a scale | 4.14 (0.10) | 3.83 (0.07) | 3.61 (0.07) | 4.39 (0.12) | 3.85 (0.08) | 3.79 (0.09)

10. Secondary Outcome: Urge to Smoke
Description: Assessed from 1=Not at all strong to 7=Extremely strong by, "How strong is your urge to smoke waterpipe tobacco right now?" Mean scores range from 1 to 7. A higher mean score reflects the participant had a stronger urge to smoke waterpipe tobacco.
Time Frame: up to 45 minutes
Population: Participants who completed the study.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Social Allure Ads Only | Social Allure Ads With Text-only Health Warning Labels (HWLs) | Social Allure Ads With Text + Graphic Health Warning Labels (HWLs) | Product Ads Only | Product Ads With Text-only Health Warning Labels (HWLs) | Product Ads With Text + Graphic Health Warning Labels (HWLs)
Number analyzed (Participants) | 300 | 602 | 598 | 201 | 402 | 401
score on a scale | 3.34 (0.12) | 3.28 (0.08) | 3.06 (0.08) | 3.82 (0.14) | 3.29 (0.10) | 3.27 (0.10)

11. Secondary Outcome: Avoidance / Acceptance of Health Warnings as Measured by Eye Tracking
Description: Participants were going to be positioned to view several ads, and with an apparatus, track their visual movements.
Time Frame: up to one hour
Population: This outcome measure required participants meeting in person with a lab researcher. However, due to COVID, where a policy was implemented on campus to not allow in-person visits for research studies, this was not possible. Hence, no data were collected and will not be collected in the future.
Arm/Group | Social Allure Ads Only | Social Allure Ads With Text-only Health Warning Labels (HWLs) | Social Allure Ads With Text + Graphic Health Warning Labels (HWLs) | Product Ads Only | Product Ads With Text-only Health Warning Labels (HWLs) | Product Ads With Text + Graphic Health Warning Labels (HWLs)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to one hour
Arm/Group | Social Allure Ads Only | Social Allure Ads With Text-only Health Warning Labels (HWLs) | Social Allure Ads With Text + Graphic Health Warning Labels (HWLs) | Product Ads Only | Product Ads With Text-only Health Warning Labels (HWLs) | Product Ads With Text + Graphic Health Warning Labels (HWLs)
All-Cause Mortality (participants affected / at risk) | 0/300 | 0/602 | 0/598 | 0/201 | 0/402 | 0/401
Serious Adverse Events (participants affected / at risk) | 0/300 | 0/602 | 0/598 | 0/201 | 0/402 | 0/401
Other Adverse Events (participants affected / at risk) | 0/300 | 0/602 | 0/598 | 0/201 | 0/402 | 0/401

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-07): https://cdn.clinicaltrials.gov/large-docs/16/NCT03723616/Prot_SAP_000.pdf